CLINICAL TRIAL: NCT06446492
Title: Impact of Video-Enhanced Consent on Informed Decision-Making for Parents of Extremely Preterm Infants Eligible for the ViDES Study: A Randomized Controlled Trial
Brief Title: Impact of Video-Enhanced Consent on Informed Decision-Making for Parents of Extremely Preterm Infants Eligible for the ViDES Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Maria del Mar Romero López, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-22-0563 (sub-study)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-12

CONDITIONS: Understanding of Consent in Clinical Research; Implementation of Video-Consent in Clinical Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video-enhanced approach to consent (Experimental): The research team will introduce themselves and ask the parents to watch an informational video explaining the ViDES study on an iPad while they stay in the room with the parents. After viewing the video, the team will answer any questions and provide written consent and enough time to decide whether to participate in the study. The research team will also provide a QR code that grants parents/guardians access to the video on their own device at any time. This allows them to pause, rewind, and revisit the information.
  Interventions: Other: ViDEO explaining study
- Usual care approach to consent (Active Comparator): The research team will present a detailed explanation of the ViDES study, answer questions, provide written consent, and provide enough time to decide on participation or not in the study.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ViDEO explaining study — The research team will introduce themselves and ask the parents to watch an informational video explaining the ViDES study on an iPad while they stay in the room with the parents. After viewing the video, the team will answer any questions and provide written consent and enough time to decide whether to participate in the study. The research team will also provide a QR code that grants parents/guardians access to the video on their own device at any time. This allows them to pause, rewind, and revisit the information.
  Arms: Video-enhanced approach to consent
Other: Usual Care — The research team will present a detailed explanation of the ViDES study, answer questions, provide written consent, and provide enough time to decide on participation or not in the study.
  Arms: Usual care approach to consent

SUMMARY:
This pilot randomized controlled trial evaluates the impact of video-enhanced consent compared to the usual approach. The investigators aim to assess if video-enhanced consent empowers decision-making and improves understanding in parents considering participation in the ViDES study, which investigates the effectiveness of Vitamin D supplementation in extremely preterm infants (the ViDES study is separately registered as NCT05459298).

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians of extremely preterm infants (<28 weeks gestational age or <1000 g birth weight) admitted to the Neonatal Intensive Care Unit at Children's Memorial Hermann hospital that qualify for the ViDES study (ViDES study is separately registered as NCT05459298)

Exclusion Criteria:

* Parents/legal guardians deaf or blind
* Parents/legal guardians unable to consent for the VIDES study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
ViDES trial consent rate | Within 1 week of the intervention
Participants' understanding of the ViDES study as assessed by a questionnaire | Within 48 hours of the intervention
  The questionnaire assesses recall of possible benefits and risks of participation.
Participants' satisfaction with consent approach as assessed by a questionnaire | Within 48 hours of the intervention
  The questionnaire assesses satisfaction with ability to ask questions and decision time.
Participant's opinions related to participation in research as assessed by a questionnaire | Within 48 hours of the intervention
  The questionnaire assesses participant's opinions related to participation in research and research being part of the care of infants.

CONTACTS AND LOCATIONS:
Overall Officials: Maria del Mar Romero López, MD, MS, PhD, Principal Investigator — The University of Texas Health Science Center at Houston (UTHealth Houston)
Locations (1):
- McGovern Medical School at UTHealth Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No